CLINICAL TRIAL: NCT02844205
Title: Evaluation of the Reproducibility of a New Practical Newborn Behavioral Observation Scale in Order to Implement an Individualized Care Program
Brief Title: Reproducibility of a New Practical Newborn Behavioral Observation Scale
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: 9589
Record Dates: First submitted 2016-07-18; First posted 2016-07-26 (Estimated); Last update posted 2016-09-01 (Estimated); Status verified 2016-08

CONDITIONS: Premature Newborn
Keywords: nursing care; observational scale; neonate; premature infant; developmental care
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: quotation of the newborn behavioral observation scale — quotation of the newborn behavioral observation scale by 12 experimented nurses. Patient will be filmed during an usual care and nurses will quote the scale thanks to the video.

SUMMARY:
Neonatal intensive care is necessary for the survival of preterm baby. Several studies show the deleterious effect on the immature brain due to stimulations caused by the environment and hospital care.

However, a specific and individualized support to the development during the first weeks of this preterm patient has a positive effect on newborn development.

A new practical newborn behavioral observation scale has been developed by the investigators care unit in order to adapt care and individualized support to the development for each patient.

The goal of this study is to estimate the external reproductibility of this scale by experimented nurse in order to implement an individualized care program.

ELIGIBILITY:
Inclusion Criteria:

* term of birth between 24 and 33 weeks of amenorrhea
* weight less than 1500g birth;
* postnatal age between 1 and 60 days
* consent form of parent in order to film their baby

Exclusion Criteria:

Ages: 1 Day to 60 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm infant hospitalized in intensive care unit.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2015-11; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
assessment of the external reproductibility of a new practical newborn behavioral observation scale | up to 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Cambonie, Professor, Principal Investigator — University Hospital, Montpellier
Locations (1):
- University hospital of Montpellier, Montpellier, France